CLINICAL TRIAL: NCT02311673
Title: A Phase 2, Randomized, Double-Blind, Placebo-controlled Pilot Study to Assess the Effects of RM-493, a Melanocortin 4 Receptor (MC4R) Agonist, in Obese Subjects With Prader-Willi Syndrome (PWS) on Safety, Weight Reduction, and Food-Related Behaviors
Brief Title: Phase 2 Trial to Evaluate Safety and Efficacy of Setmelanotide (RM-493) in Obese Participants With Prader-Willi Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM-493-010; R01FD005094-01A1 (FDA)
Record Dates: First submitted 2014-11-25; First posted 2014-12-08 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome; obesity; hyperphagia
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity; Hyperphagia | interventions — setmelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Setmelanotide 0.5 mg (Experimental): Participants received setmelanotide 0.5 milligrams (mg) once daily as a subcutaneous injection from Day 15 to Day 41 (4-week, double-blind randomized treatment period) and Day 42 to Day 55 (2-week, randomized withdrawal period).
  Interventions: Drug: Setmelanotide
- Setmelanotide 1.5 mg (Experimental): Participants received setmelanotide 1.5 once daily as a subcutaneous injection from Day 15 to Day 41 (4-week, double-blind randomized treatment period), Day 42 to Day 55 (2-week, randomized withdrawal period), and Day 56 to Day 69 (optional 2-week, open-label extension period).
  Interventions: Drug: Setmelanotide
- Setmelanotide 2.5 mg (Experimental): Participants received setmelanotide 2.5 once daily as a subcutaneous injection from Day 15 to Day 41 (4-week, double-blind randomized treatment period), Day 42 to Day 55 (2-week, randomized withdrawal period), and Day 56 to Day 69 (optional 2-week, open-label extension period).
  Interventions: Drug: Setmelanotide
- Placebo (Placebo Comparator): Participants received placebo matched to setmelanotide once daily as a subcutaneous injection from Day 1 to Day 14 (2-week, single-blind run-in period), Day 15 to Day 41 (4-week, double-blind randomized treatment period), and Day 42 to Day 55 (2-week, randomized withdrawal period).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Setmelanotide — subcutaneous injection
  Other Names: RM-493
  Arms: Setmelanotide 0.5 mg; Setmelanotide 1.5 mg; Setmelanotide 2.5 mg
Drug: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the effects of a once daily subcutaneous injectable formulation of setmelanotide in obese participants with Prader-Willi syndrome on tolerability, weight loss, and hyperphagia-related behavior. The study drug (setmelanotide and placebo) was administered in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

1. PWS due to chromosome 15 micro-deletion, maternal uniparental disomy, or imprinting defect, confirmed by fluorescent in situ hybridization, chromosomal microarray, and/or methylation studies. Obese male or female participants weighing at least 50 kilograms (kg) with body mass index (BMI) ≥ 27 kilogram per square meter (kg/m²)
2. Age 16-65 years
3. If a participant has diagnosis of type 2 diabetes, following criteria must be met:

   1. hemoglobin A1C (HbA1c) < 7.5% not being managed with insulin. Participants taking glucagon-like peptide-1 (GLP-1) analogues (exenatide or liraglutide) must have been on stable dose for greater than 3 months.
   2. Fasting plasma glucose < 140 milligrams per deciliter (mg/dL)
   3. No history of ketoacidosis or hyperosmolar coma
4. Vital signs must be within the following ranges and stable.

   1. Systolic blood pressure, 90-150 millimeter of mercury (mm Hg)
   2. Diastolic blood pressure, 50-90 mm Hg
   3. Pulse rate, 40-100 beats per minute (bpm)
5. Stable body weight at home for approximately 2 months (self or guardian-reported loss/gain within ± 5%).
6. Blood pressure (≤ 150/90 mmHg); may include stable dose (≥ 30 days of use) of up to two anti-hypertensive medications that are intended to remain on a stable dose during the protocol
7. Parent or guardian is able to communicate well with the investigator, to understand and comply with the requirements of the study, and be able to understand and sign the written informed consent. Due to the significant intellectual disability with PWS, assent is to be provided by the participant who cannot consent for himself or herself.
8. Results of screening clinical laboratory tests (complete blood count with differential and platelets and chemistry profile) must be within normal range or, if outside of the normal range, must be accepted by the investigator and sponsor as not clinically significant.
9. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months (and confirmed with a screening follicle-stimulating hormone (FSH) level in the post-menopausal lab range), do not require contraception during the study. All other females of child-bearing potential must agree to use contraception as outlined in the protocol.
10. Males with female partners of childbearing potential must agree to a double barrier method if they become sexually active during the study and for 90 days following the study. Male participants must not donate sperm for 90 days following their participation in the study.
11. Participants must be on a stable dose of any allowed chronic concomitant medications while participating in the study.

Exclusion Criteria:

1. Recent use (within 3 month) of weight loss agents including herbal medication.
2. Diagnosis of schizophrenia, bipolar disorder, personality disorder or other Diagnostic and Statistical Manual of Mental Disorders, Third Edition (DSM-III) disorders which the investigator believes will interfere significantly with study compliance.
3. A Patient Health Questionnaire-9 (PHQ-9) score of ≥ 15.
4. Any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS).
5. Clinically significant illness in the 8 weeks before screening.
6. History of clinically significant bleeding disorders.
7. Current, clinically significant liver, renal, pulmonary, cardiac, oncologic, or gastrointestinal disease.
8. Diagnosis of type 1 diabetes mellitus or other active endocrine disorders (e.g., Cushing syndrome, or thyroid dysfunction except if on adequate thyroid or glucocorticoid replacement supplement).
9. Cardiovascular disease event including history of congestive heart failure, coronary artery disease, myocardial infarction, second degree or greater heart block or prolonged QT syndrome.
10. Blood pressure > 150/90 mm Hg.
11. Liver disease or liver injury as indicated by abnormal liver function tests, aspartate aminotransferase, alkaline phosphatase, or serum bilirubin (> 1.5 x upper limit of normal for any of these tests) or history of hepatic cirrhosis.
12. History or presence of impaired renal function as indicated by clinically significantly abnormal creatinine, blood urea nitrogen, or urinary constituents (e.g., albuminuria) or moderate to severe renal dysfunction as defined by the Cockcroft-Gault equation (< 50 mL/min).
13. History or close family history (parents or siblings) of melanoma.
14. Oculocutaneous albinism (occurs at approximately 1% in PWS).
15. Significant dermatologic findings as part of the Screening comprehensive skin evaluation performed by the dermatologist.
16. Significant history of abuse of drugs or solvents in the year before screening or a positive Drugs of Abuse (DOA) test at screening.
17. History of alcohol abuse in the past year before screening or currently drinks in excess of 21 units per week (3 servings or units/day).
18. Caffeine consumption exceeding 6 cups of caffeinated tea/coffee (or equivalent) per day.
19. Participant is, in the opinion of the Investigator, not suitable to participate in the study.
20. Participation in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing.
21. Positive history for human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C tests or tuberculosis.
22. Serious adverse reaction or significant hypersensitivity to any drug.
23. Clinically significant blood loss or blood donation > 500 milliliters (mL) within 3 months.
24. Inadequate venous access.
25. History of low blood counts or recurring infections.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2016-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, Study Director — Rhythm Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - University of California Irvine, Irvine, California
  - University of Florida, Gainesville, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - Winthrop University Hospital, Mineola, New York
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 44 participants screened, 40 participants were enrolled in the study.
Groups:
- Setmelanotide 0.5 mg: Participants received placebo matched to setmelanotide once daily as a subcutaneous injection from Day 1 to Day 14 (2-week, single-blind placebo run-in period); thereafter, participants received setmelanotide 0.5 milligrams (mg) once daily as a subcutaneous injection from Day 15 to Day 41 (4-week, double-blind randomized treatment period) and Day 42 to Day 55 (2-week, randomized withdrawal period).
- Setmelanotide 1.5 mg: Participants received placebo matched to setmelanotide once daily as a subcutaneous injection from Day 1 to Day 14 (2-week, single-blind placebo run-in period); thereafter, participants received setmelanotide 1.5 once daily as a subcutaneous injection from Day 15 to Day 41 (4-week, double-blind randomized treatment period), Day 42 to Day 55 (2-week, randomized withdrawal period), and Day 56 to Day 69 (optional 2-week, open-label extension period).
- Setmelanotide 2.5 mg: Participants received placebo matched to setmelanotide once daily as a subcutaneous injection from Day 1 to Day 14 (2-week, single-blind placebo run-in period); thereafter, participants received setmelanotide 2.5 once daily as a subcutaneous injection from Day 15 to Day 41 (4-week, double-blind randomized treatment period), Day 42 to Day 55 (2-week, randomized withdrawal period), and Day 56 to Day 69 (optional 2-week, open-label extension period).
- Placebo: Participants received placebo matched to setmelanotide once daily as a subcutaneous injection from Day 1 to Day 14 (2-week, single-blind placebo run-in period), Day 15 to Day 41 (4-week, double-blind randomized treatment period), and Day 42 to Day 55 (2-week, randomized withdrawal period).
Period: Placebo Run-in Period 1 (2 Weeks)
Arm/Group | Setmelanotide 0.5 mg | Setmelanotide 1.5 mg | Setmelanotide 2.5 mg | Placebo
Started | 0 | 0 | 0 | 40
Completed | 0 | 0 | 0 | 40
Not Completed | 0 | 0 | 0 | 0
Period: Double-blind Randomized Period 2 (4 Wks)
Arm/Group | Setmelanotide 0.5 mg | Setmelanotide 1.5 mg | Setmelanotide 2.5 mg | Placebo
Started (Forty participants who completed placebo single-blind run-in period entered the double-blind randomized treatment period. Fifteen participants continued placebo and 25 participants were randomized to other treatment groups in the double-blind randomized treatment period.) | 4 | 13 (One participant was randomized to setmelanotide 2.5 mg treatment group and treated with setmelanotide 1.5 mg group.) | 8 | 15 (One participant was randomized to setmelanotide 2.5 mg treatment group and treated with placebo.)
Completed | 4 | 13 | 7 | 15
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by participant and Investigator decision | 0 | 0 | 1 | 0
Period: Randomized Withdrawal Period 3 (2 Weeks)
Arm/Group | Setmelanotide 0.5 mg | Setmelanotide 1.5 mg | Setmelanotide 2.5 mg | Placebo
Started (After completion of Period 2, a randomized withdrawal (Period 3) was initiated; participants within each of the setmelanotide groups were randomized 1:1; participants who had received setmelanotide were either continued at the current active dose, or switched to placebo treatment. Participants administered placebo during Period 2 were randomized 1:1 in Period 3 and either continued to receive placebo or began to receive setmelanotide.) | 3 | 10 | 5 | 20
Completed | 3 | 10 | 5 | 20
Not Completed | 0 | 0 | 0 | 0
Period: Open-label Extension Period 4 (2 Weeks)
Arm/Group | Setmelanotide 0.5 mg | Setmelanotide 1.5 mg | Setmelanotide 2.5 mg | Placebo
Started (Period 4 was a follow-up, open-label extension available to participants who completed the first 3 periods and wanted to continue treatment. In Period 4, all participants were to receive either setmelanotide 1.5 mg or setmelanotide 2.5 mg.) | 0 | 22 (Three participants were randomized to setmelanotide 2.5 mg treatment group and treated with setmelanotide 1.5 mg.) | 16 | 1 (One participant advanced from the Double-blind Randomized Treatment Period (Period 2) to the Open-Label Extension Period (Period 4) due to an error in the interactive voice response system (IVRS); therefore, results are presented for 38 participants in Randomized Withdrawal Period (Period 3) but 39 participants in the Open-Label Extension Period (Period 4). The participant was randomized to setmelanotide 2.5 mg treatment group and treated with placebo.)
Completed | 0 | 22 | 16 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all randomized participants who received at least 1 dose of study medication, and had at least one post-dose safety assessment (within Period 2). Participants were classified into groups based on actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Setmelanotide 0.5 mg | Setmelanotide 1.5 mg | Setmelanotide 2.5 mg | Placebo | Total
Number analyzed (Participants) | 4 | 13 | 8 | 15 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (4.19) | 24.1 (5.42) | 25.0 (9.62) | 30.5 (11.97) | 26.4 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 6 | 7 | 21
  Male | 2 | 7 | 2 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 1 | 4
  Not Hispanic or Latino | 2 | 13 | 7 | 14 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 4 | 9 | 8 | 15 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Treatment-Emergent Adverse Event (TEAE) - Period 2
Description: An adverse event (AE) was any untoward medical occurrence in a clinical trial participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE is considered to be treatment-emergent if the onset date/time is during or after administration of double-blind study drug or, in the event that onset time precedes double-blind study drug administration, the AE increases in severity during or after administration of double-blind study drug; in either case through 1-week after the last treatment dose. A serious adverse event (SAE) was any untoward medical occurrence that, at any dose:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent disability/incapacity;
  * Was a congenital anomaly/birth defect
Time Frame: Days 15 to 41
Population: Safety Set. Participants were classified into groups based on actual treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Setmelanotide 0.5 mg (Double-blind Randomized Treatment): Participants received setmelanotide 0.5 mg once daily from Day 15 to Day 41 as a subcutaneous injection in a 4-week, double-blind randomized treatment period.
- Setmelanotide 1.5 mg (Double-blind Randomized Treatment): Participants received setmelanotide 1.5 mg once daily from Day 15 to Day 41 as a subcutaneous injection in a 4-week, double-blind randomized treatment period.
- Setmelanotide 2.5 mg (Double-blind Randomized Treatment): Participants received setmelanotide 2.5 mg once daily from Day 15 to Day 41 as a subcutaneous injection in a 4-week, double-blind randomized treatment period.
- Placebo (Double-blind Randomized Treatment): Participants received placebo matched to setmelanotide once daily from Day 15 to Day 41 as a subcutaneous injection in a 4-week, double-blind randomized treatment period.
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 13 | 8 | 15
Participants
  Participants with at least 1 TEAE | 4 | 11 | 6 | 11
  Participants with at least 1 SAE | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced a TEAE - Period 3
Description: An AE was any untoward medical occurrence in a clinical trial participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE is considered to be treatment-emergent if the onset date/time is during or after administration of double-blind study drug or, in the event that onset time precedes double-blind study drug administration, the AE increases in severity during or after administration of double-blind study drug; in either case through 1-week after the last treatment dose. An SAE was any untoward medical occurrence that, at any dose:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent disability/incapacity;
  * Was a congenital anomaly/birth defect
Time Frame: Days 42 to 55
Population: Participants in the Safety Set with available data were analyzed. Participants were classified into groups based on actual treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Setmelanotide 0.5 mg (Randomized Withdrawal Period): Participants received setmelanotide 0.5 mg once daily from Day 42 to Day 55 as a subcutaneous injection in a 2-week, randomized withdrawal period.
- Setmelanotide 1.5 mg (Randomized Withdrawal Period): Participants received setmelanotide 1.5 mg once daily from Day 42 to Day 55 as a subcutaneous injection in a 2-week, randomized withdrawal period.
- Setmelanotide 2.5 mg (Randomized Withdrawal Period): Participants received setmelanotide 2.5 mg once daily from Day 42 to Day 55 as a subcutaneous injection in a 2-week, randomized withdrawal period.
- Placebo (Randomized Withdrawal Period): Participants received placebo matched to setmelanotide once daily from Day 42 to Day 55 as a subcutaneous injection in a 2-week, randomized withdrawal period.
Arm/Group | Setmelanotide 0.5 mg (Randomized Withdrawal Period) | Setmelanotide 1.5 mg (Randomized Withdrawal Period) | Setmelanotide 2.5 mg (Randomized Withdrawal Period) | Placebo (Randomized Withdrawal Period)
Number analyzed (Participants) | 3 | 10 | 5 | 20
Participants
  Participants with at least 1 TEAE | 3 | 7 | 4 | 11
  Participants with at least 1 SAE | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced a TEAE - Period 4
Description: as for outcome 2
Time Frame: Days 56 to 69
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Setmelanotide 1.5 mg (Open-Label Extension): Participants received setmelanotide 1.5 mg once daily from Day 56 to Day 69 as a subcutaneous injection in an optional 2-week, open-label extension period.
- Setmelanotide 2.5 mg (Open-Label Extension): Participants received setmelanotide 2.5 mg once daily from Day 56 to Day 69 as a subcutaneous injection in an optional 2-week, open-label extension period.
- Placebo (Open-Label Extension): Participants received placebo matched to setmelanotide once daily from Day 56 to Day 69 as a subcutaneous injection in an optional 2-week, open-label extension period.
Arm/Group | Setmelanotide 1.5 mg (Open-Label Extension) | Setmelanotide 2.5 mg (Open-Label Extension) | Placebo (Open-Label Extension)
Number analyzed (Participants) | 22 | 16 | 1
Participants
  Participants with at least 1 TEAE | 17 | 12 | 0
  Participants with at least 1 SAE | 0 | 0 | 0

4. Primary Outcome: Mean Body Weight - Period 2
Time Frame: Baseline (Day 15)
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of randomized study medication with a baseline and at least 1 postbaseline efficacy observation within Period 2. Participants were classified based on randomized treatment group, regardless of the actual treatment received. Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 12 | 9 | 13
Kilograms (kg) | 94.3 (16.84) | 92.7 (5.50) | 101.6 (5.35) | 102.2 (9.16)

5. Primary Outcome: Percent Change From Baseline in Body Weight - Period 2
Time Frame: Baseline (Day 15) and Day 42
Population: Participants in the FAS with available data were analyzed. Participants were classified based on randomized treatment group, regardless of the actual treatment received.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 12 | 9 | 13
percent change | -0.7 [-3.1 to 1.8] | -0.8 [-2.2 to 0.6] | 0.4 [-1.2 to 2.0] | -0.4 [-1.8 to 0.9]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.420, Longitudinal mixed analysis of variance — One sided p-value; Least Squares (LS) Mean Difference = -0.3, 95% CI 2-sided [-3.1 to 2.5] — A longitudinal mixed analysis of variance model with fixed effects for treatment, time, treatment-by-time interaction, treatment-by-baseline weight interaction, baseline weight as covariate and participant as random effect was used
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.348, Longitudinal mixed analysis of variance; One sided p-value; LS Mean Difference = -0.4, 95% CI 2-sided [-2.3 to 1.6] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.779, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 0.8, 95% CI 2-sided [-1.3 to 2.9] — [estimate comment as in outcome 5, analysis 1]

6. Primary Outcome: Overall Score of Prader-Willi Syndrome (PWS) Hyperphagia Questionnaire - Period 2
Description: The hyperphagia questionnaire is a 10-item instrument designed to measure food-related preoccupations and problems in PWS, as well as the severity of these concerns. Three factors identified from this questionnaire are: Hyperphagic Drive, Hyperphagic Behaviors, and Hyperphagic Severity. Items are rated by care providers on a 5-point scale (1=not a problem to 5=a severe and/or frequent problem). Raw scores for each factor were used in data analyses, and the 3 domains were summed for an overall summary index of hyperphagia. Possible scores on the questionnaire range from a minimum score of 10 (no hyperphagia) to a maximum score of 50 (greater hyperphagia).
Time Frame: Baseline (Day 15)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 12 | 9 | 13
units on a scale | 31.0 (2.86) | 21.2 (2.28) | 20.2 (2.79) | 18.7 (2.33)

7. Primary Outcome: Percent Change From Baseline in Overall Score of Prader-Willi Syndrome (PWS) Hyperphagia Questionnaire - Period 2
Description: The hyperphagia questionnaire is a 10-item instrument designed to measure food-related preoccupations and problems in PWS, as well as the severity of these concerns. Three factors identified from this questionnaire are: Hyperphagic Drive, Hyperphagic Behaviors, and Hyperphagic Severity. Items are rated by care providers on a 5-point scale (1=not a problem to 5=a severe and/or frequent problem). Raw scores for each factor were used in data analyses, and the 3 domains were summed for an overall summary index of hyperphagia. Possible scores on the questionnaire range from a minimum score of 10 (no hyperphagia) to a maximum score of 50 (greater hyperphagia). Percent change from baseline in overall score of PWS hyperphagia questionnaire is presented.
Time Frame: Baseline (Day 15) and Day 42
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 12 | 9 | 13
percent change | 20.2 [-8.7 to 49.1] | -5.2 [-21.3 to 10.9] | -5.0 [-23.7 to 13.6] | -1.3 [-16.9 to 14.3]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.901, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 21.5, 95% CI 2-sided [-11.8 to 54.8] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.362, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -3.9, 95% CI 2-sided [-26.3 to 18.5] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.378, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -3.7, 95% CI 2-sided [-28.0 to 20.5] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Percent Change From Baseline in Hyperphagic Drive Score of PWS Hyperphagia Questionnaire - Period 2
Description: The hyperphagia questionnaire is a 10-item instrument designed to measure food-related preoccupations and problems in PWS, as well as the severity of these concerns. Hyperphagic drive score assesses the persistence in asking for food based on 4 items. All 4 items are rated by care providers on a 5-point scale (1=not a problem to 5=a severe and/or frequent problem). Possible scores for hyperphagic drive range from a minimum score of 4 (no hyperphagic drive) to a maximum score of 20 (greater hyperphagic drive). Percent change from baseline in hyperphagic drive score of PWS hyperphagia questionnaire is presented.
Time Frame: Baseline (Day 15) and Day 42
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 12 | 9 | 13
percent change | 27.2 [-8.9 to 63.3] | -3.6 [-24.1 to 16.9] | -6.8 [-30.5 to 16.8] | 6.6 [-13.2 to 26.4]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.840, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 20.6, 95% CI 2-sided [-20.9 to 62.2] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.236, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -10.2, 95% CI 2-sided [-38.7 to 18.4] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.191, Longitudinal mixed analysis of variance; One sided p-value; LS Mean Difference = -13.4, 95% CI 2-sided [-44.2 to 17.4]

9. Secondary Outcome: Percent Change From Baseline in Hyperphagic Behaviors Score of PWS Hyperphagia Questionnaire - Period 2
Description: The hyperphagia questionnaire is a 10-item instrument designed to measure food-related preoccupations and problems in PWS, as well as the severity of these concerns. Hyperphagic behavior factor score assesses food seeking behaviors based on 4 items. All 4 items are rated by care providers on a 5-point scale (1=not a problem to 5=a severe and/or frequent problem). Possible scores for hyperphagic behaviors range from a minimum score of 4 (no hyperphagic behavior) to a maximum score of 20 (greater hyperphagic behavior). Percent change from baseline in hyperphagic behaviors score of PWS hyperphagia questionnaire is presented.
Time Frame: Baseline (Day 15) and Day 42
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 12 | 9 | 13
percent change | 19.1 [-19.3 to 57.5] | -1.7 [-22.3 to 18.9] | -3.0 [-26.8 to 20.8] | -0.4 [-20.4 to 19.6]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.812, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 19.5, 95% CI 2-sided [-24.8 to 63.8]; A longitudinal mixed analysis of variance model with fixed effects for treatment, time, treatment-by-time interaction, treatment-by-baseline weight interaction, baseline weight as covariate and participant as random effect was used
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.464, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -1.3, 95% CI 2-sided [-29.9 to 27.4] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.432, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -2.6, 95% CI 2-sided [-33.6 to 28.4] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Percent Change From Baseline in Hyperphagic Severity Score of PWS Hyperphagia Questionnaire - Period 2
Description: The hyperphagia questionnaire is a 10-item instrument designed to measure food-related preoccupations and problems in PWS, as well as the severity of these concerns. Hyperphagic severity factor score assesses the severity of hyperphagia based on 2 items. Both items are rated by care providers on a 5-point scale (1=not a problem to 5=a severe and/or frequent problem). Possible scores for hyperphagic severity range from a minimum score of 2 (no hyperphagic severity) to a maximum score of 10 (greater hyperphagic severity). Percent change from baseline in hyperphagic severity score of PWS hyperphagia questionnaire is presented.
Time Frame: Baseline (Day 15) and Day 42
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 12 | 9 | 13
percent change | 33.2 [-4.4 to 70.9] | -0.7 [-22.1 to 20.6] | 5.5 [-19.1 to 30.2] | -16.7 [-37.3 to 3.9]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.988, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 49.9, 95% CI 2-sided [6.7 to 93.2] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.859, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 16.0, 95% CI 2-sided [-13.7 to 45.6] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.916, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 22.2, 95% CI 2-sided [-9.8 to 54.3] — [estimate comment as in outcome 5, analysis 1]

11. Secondary Outcome: Percent Change From Baseline in Overall Score of PWS Hyperphagia Questionnaire - Period 3
Description: as for outcome 7
Time Frame: Baseline (Day 42) and Day 56
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Setmelanotide 0.5 mg (Randomized Withdrawal Period) | Setmelanotide 1.5 mg (Randomized Withdrawal Period) | Setmelanotide 2.5 mg (Randomized Withdrawal Period) | Placebo (Randomized Withdrawal Period)
Number analyzed (Participants) | 3 | 10 | 5 | 20
percent change | 35.0 [-2.9 to 72.9] | -1.8 [-18.4 to 14.7] | 3.4 [-20.1 to 26.9] | 2.3 [-9.6 to 14.2]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Randomized Withdrawal Period) vs Placebo (Randomized Withdrawal Period); Test type: Other; p = 0.943, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 32.7, 95% CI 2-sided [-8.4 to 73.8] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Randomized Withdrawal Period) vs Placebo (Randomized Withdrawal Period); Test type: Other; p = 0.339, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -4.2, 95% CI 2-sided [-24.4 to 16.1] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Randomized Withdrawal Period) vs Placebo (Randomized Withdrawal Period); Test type: Other; p = 0.533, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 1.1, 95% CI 2-sided [-25.0 to 27.2] — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Percent Change From Baseline in Overall Score of PWS Hyperphagia Questionnaire - Period 4
Description: as for outcome 7
Time Frame: Baseline (Day 56) and Day 70
Population: Participants in the FAS with available data were analyzed. In Period 4, one participant was randomized to setmelanotide 2.5 mg treatment group but treated with placebo. As participants in the FAS are classified based on randomized treatment group regardless of the actual treatment received, the placebo group is not included in the FAS analysis for Period 4.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Setmelanotide 1.5 mg (Open-Label Extension) | Setmelanotide 2.5 mg (Open-Label Extension)
Number analyzed (Participants) | 15 | 20
percent change | -0.9 (23.21) | -0.4 (29.94)

13. Secondary Outcome: Mean Setmelanotide Trough Concentrations
Description: The average of setmelanotide trough concentrations values for both timepoints (5 minutes predose on Day 42 and Day 70) is presented.
Time Frame: 5 minutes predose on Day 42 and Day 70
Population: The Pharmacokinetic (PK) Evaluable Population was defined as all participants in the Safety Population who had evaluable plasma concentration-time profiles for setmelanotide in the substudy. One participant may have received more than one doses in different periods (eg, 0.5 mg in the Double-blind Randomized Treatment Period and 1.5 mg in the Randomized Withdrawal Period) and therefore included in multiple groups in the data presented.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Setmelanotide 0.5 mg: Participants received setmelanotide 0.5 mg once daily as a subcutaneous injection from Day 15 to Day 41 (4-week, double-blind randomized treatment period) and Day 42 to Day 55 (2-week, randomized withdrawal period).
Arm/Group | Setmelanotide 0.5 mg | Setmelanotide 1.5 mg | Setmelanotide 2.5 mg
Number analyzed (Participants) | 4 | 27 | 29
nanograms per milliliter (ng/mL) | 0.790 (0.336) | 2.59 (1.51) | 5.63 (4.19)

14. Secondary Outcome: Maximum Drug Concentration (Cmax) of Setmelanotide During a 24-Hour Steady-State Interval
Description: Maximum drug concentration determined directly from individual concentration-time data.
Time Frame: Starting on any day from Day 63 through 69, a 24-hour PK profile obtained; blood samples were collected at 0 (within 5 minutes predose), 1, 2, 4, 6, 7, 8, 9, 10, 12, and 24 hours after dosing
Population: Participants in the PK Evaluable Population with available data were analyzed. Because only 1 participant was analyzed in the setmelanotide 1.5 mg group, no data are reported for this group in order to protect and maintain participant privacy/confidentiality.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Setmelanotide 2.5 mg (Open-Label Extension)
Number analyzed (Participants) | 7
ng/mL | 39.1 (12.2)

15. Secondary Outcome: Time to the Maximum Drug Concentration (Tmax) of Setmelanotide During a 24-Hour Steady-State Interval
Description: Maximum drug concentration determined directly from individual concentration-time data.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Setmelanotide 2.5 mg (Open-Label Extension)
Number analyzed (Participants) | 7
hours (hr) | 6.00 [5.95 to 10.15]

16. Secondary Outcome: Area Under the Drug Concentration-Time Curve From Time-Zero to 24 Hours Postdose (AUC24h) of Setmelanotide During a 24-Hour Steady-State Interval
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Setmelanotide 2.5 mg (Open-Label Extension)
Number analyzed (Participants) | 5
hr*ng/mL | 569.4 (190.6)

17. Secondary Outcome: Volume of Distribution (Vd) of Setmelanotide During a 24-Hour Steady-State Interval
Description: Volume of distribution calculated as Dose/The observed terminal rate constant*AUC24h.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Setmelanotide 2.5 mg (Open-Label Extension)
Number analyzed (Participants) | 5
Liters (L) | 52.8 (10.0)

18. Secondary Outcome: Total Clearance (CL) of Setmelanotide During a 24-Hour Steady-State Interval
Description: Clearance after extravascular administration; calculated as Dose/AUC24h.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Setmelanotide 2.5 mg (Open-Label Extension)
Number analyzed (Participants) | 5
L/hr | 4.77 (1.49)

19. Secondary Outcome: Change From Baseline in Body Weight - Period 2
Time Frame: Baseline (Day 15) and Day 42
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 12 | 9 | 13
kg | -0.6 [-3.1 to 1.8] | -0.8 [-2.2 to 0.7] | 0.3 [-1.4 to 1.9] | -0.4 [-1.8 to 1.0]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.439, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -0.2, 95% CI 2-sided [-3.0 to 2.6] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.366, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -0.3, 95% CI 2-sided [-2.3 to 1.6] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.744, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 0.7, 95% CI 2-sided [-1.4 to 2.8] — [estimate comment as in outcome 5, analysis 1]

20. Secondary Outcome: Percent Change From Baseline in Body Weight - Period 3
Time Frame: Baseline (Day 42) and Day 56
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Setmelanotide 0.5 mg (Randomized Withdrawal Period) | Setmelanotide 1.5 mg (Randomized Withdrawal Period) | Setmelanotide 2.5 mg (Randomized Withdrawal Period) | Placebo (Randomized Withdrawal Period)
Number analyzed (Participants) | 3 | 10 | 5 | 20
percent change | 1.3 [-0.3 to 2.9] | 0.0 [-0.9 to 0.9] | 0.0 [-1.3 to 1.3] | 0.2 [-0.4 to 0.9]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Randomized Withdrawal Period) vs Placebo (Randomized Withdrawal Period); Test type: Other; p = 0.883, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 1.0, 95% CI 2-sided [-0.7 to 2.8] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Randomized Withdrawal Period) vs Placebo (Randomized Withdrawal Period); Test type: Other; p = 0.338, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -0.2, 95% CI 2-sided [-1.3 to 0.9] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Randomized Withdrawal Period) vs Placebo (Randomized Withdrawal Period); Test type: Other; p = 0.381, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -0.2, 95% CI 2-sided [-1.6 to 1.2] — [estimate comment as in outcome 5, analysis 1]

21. Secondary Outcome: Percent Change From Baseline in Body Weight - Period 4
Time Frame: Baseline (Day 56) and Day 70
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Setmelanotide 1.5 mg (Open-Label Extension) | Setmelanotide 2.5 mg (Open-Label Extension)
Number analyzed (Participants) | 19 | 20
percent change | -0.0 (0.90) | 0.0 (2.70)

22. Secondary Outcome: Percent Change From Baseline in Body Weight for Continuous Active and Continuous Placebo Treatments - Period 2 and 3
Time Frame: Baseline (Day 15), Day 42, Day 56
Population: FAS population with available data were analyzed for participants who continued with the same treatment when switched from Double-blind Randomized Treatment to Randomized Withdrawal Period.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Setmelanotide 0.5 mg (Double-blind Randomized Treatment, Then Randomized Withdrawal Period): Participants received setmelanotide 0.5 mg as a subcutaneous injection once daily from Day 15 to Day 41 in a 4-week, double-blind randomized treatment period and then from Day 42 to Day 55 in a 2-week, randomized withdrawal period.
- Setmelanotide 1.5 mg (Double-blind Randomized Treatment, Then Randomized Withdrawal Period): Participants received setmelanotide 1.5 mg as a subcutaneous injection once daily from Day 15 to Day 41 in a 4-week, double-blind randomized treatment period and then from Day 42 to Day 55 in a 2-week, randomized withdrawal period.
- Setmelanotide 2.5 mg (Double-blind Randomized Treatment, Then Randomized Withdrawal Period): Participants received setmelanotide 2.5 mg as a subcutaneous injection once daily from Day 15 to Day 41 in a 4-week, double-blind randomized treatment period and then from Day 42 to Day 55 in a 2-week, randomized withdrawal period.
- Placebo (Double-blind Randomized Treatment), Then Placebo (Randomized Withdrawal Period): Participants received placebo matched to setmelanotide as a subcutaneous injection once daily from Day 15 to Day 41 in a 4-week, double-blind randomized treatment period and then from Day 42 to Day 55 in a 2-week, randomized withdrawal period.
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment, Then Randomized Withdrawal Period) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment, Then Randomized Withdrawal Period) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment, Then Randomized Withdrawal Period) | Placebo (Double-blind Randomized Treatment), Then Placebo (Randomized Withdrawal Period)
Number analyzed (Participants) | 2 | 6 | 4 | 7
percent change
  Percent change at Day 42 | -0.7 [-5.3 to 3.9] | -0.5 [-3.1 to 2.2] | 0.7 [-2.6 to 4.0] | -0.7 [-3.2 to 1.7]
  Percent change at Day 56 | 0.2 [-4.8 to 5.3] | -0.4 [-3.3 to 2.6] | 0.9 [-2.7 to 4.4] | -1.0 [-3.8 to 1.7]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Double-blind Randomized Treatment, Then Randomized Withdrawal Period) vs Placebo (Double-blind Randomized Treatment), Then Placebo (Randomized Withdrawal Period); Statistical analysis is provided for percent change from baseline at Day 56; Test type: Other; p = 0.679, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 1.3, 95% CI 2-sided [-4.5 to 7.0] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Double-blind Randomized Treatment, Then Randomized Withdrawal Period) vs Placebo (Double-blind Randomized Treatment), Then Placebo (Randomized Withdrawal Period); Statistical analysis is provided for percent change from baseline at Day 56; Test type: Other; p = 0.641, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 0.7, 95% CI 2-sided [-3.3 to 4.7] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Double-blind Randomized Treatment, Then Randomized Withdrawal Period) vs Placebo (Double-blind Randomized Treatment), Then Placebo (Randomized Withdrawal Period); Statistical analysis is provided for percent change from baseline at Day 56; Test type: Other; p = 0.809, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 1.9, 95% CI 2-sided [-2.6 to 6.4] — [estimate comment as in outcome 5, analysis 1]

23. Secondary Outcome: Percent Change From Baseline in Body Fat Measured Using Dual x-Ray Absorptiometry (DEXA) - Period 2
Description: Total body fat was assessed by DEXA scan.
Time Frame: Baseline (Day 15) and Day 42
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 12 | 8 | 13
percent change | -0.6 [-3.4 to 2.1] | -1.1 [-2.7 to 0.5] | -0.7 [-2.6 to 1.3] | -1.1 [-2.7 to 0.4]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.633, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 0.5, 95% CI 2-sided [-2.6 to 3.6] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.528, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 0.1, 95% CI 2-sided [-2.1 to 2.3] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.648, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 0.5, 95% CI 2-sided [-2.0 to 2.9] — [estimate comment as in outcome 5, analysis 1]

24. Secondary Outcome: Number of Participants With Clinically Significant Percent Change From Baseline in Body Fat Measured Using DEXA - Period 4
Description: Total body fat was assessed by DEXA scan. Number of participants with clinically significant percent change from baseline in body fat were judged by investigator.
Time Frame: Baseline (Day 56) and Day 70
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Setmelanotide 1.5 mg (Open-Label Extension) | Setmelanotide 2.5 mg (Open-Label Extension)
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0

25. Secondary Outcome: Percent Change From Baseline in Body Mass Measured Using DEXA - Period 2
Description: Total body mass was assessed by DEXA scan.
Time Frame: Baseline (Day 15) and Day 42
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment)
Number analyzed (Participants) | 4 | 12 | 8 | 13
percent change | -0.2 [-2.3 to 1.9] | -1.1 [-2.3 to 0.2] | -0.3 [-1.8 to 1.2] | -0.9 [-2.1 to 0.3]
Statistical Analysis 1: Comparison: Setmelanotide 0.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.712, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 0.7, 95% CI 2-sided [-1.8 to 3.1] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Setmelanotide 1.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.414, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -0.2, 95% CI 2-sided [-1.9 to 1.5] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Setmelanotide 2.5 mg (Double-blind Randomized Treatment) vs Placebo (Double-blind Randomized Treatment); Test type: Other; p = 0.732, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = 0.6, 95% CI 2-sided [-1.3 to 2.5] — [estimate comment as in outcome 5, analysis 1]

26. Secondary Outcome: Number of Participants With Clinically Significant Percent Change From Baseline in Body Mass Measured Using DEXA - Period 4
Description: Total body mass was assessed by DEXA scan. Number of participants with clinically significant percent change from baseline in body mass were judged by investigator.
Time Frame: Baseline (Day 56) and Day 70
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Setmelanotide 1.5 mg (Open-Label Extension) | Setmelanotide 2.5 mg (Open-Label Extension)
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 15 to Day 69
Description: Safety Set; participants were classified into groups based on actual treatment received. The single-blind placebo run-in period (Day 1 to Day 14) is not part of statistical analysis of this study; therefore, no AE data were collected for this period.
Groups:
- Placebo (Open-Label Extension): The participant, due to an error in the IVRS, received placebo matched to setmelanotide once daily from Day 56 to Day 69 as a subcutaneous injection in an optional 2-week, open-label extension period.
Arm/Group | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) | Placebo (Double-blind Randomized Treatment) | Setmelanotide 0.5 mg (Randomized Withdrawal Period) | Setmelanotide 1.5 mg (Randomized Withdrawal Period) | Setmelanotide 2.5 mg (Randomized Withdrawal Period) | Placebo (Randomized Withdrawal Period) | Setmelanotide 1.5 mg (Open-Label Extension) | Setmelanotide 2.5 mg (Open-Label Extension) | Placebo (Open-Label Extension)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/13 | 0/8 | 0/15 | 0/3 | 0/10 | 0/5 | 0/20 | 0/22 | 0/16 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/13 | 0/8 | 0/15 | 0/3 | 0/10 | 0/5 | 0/20 | 0/22 | 0/16 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 11/13 | 6/8 | 11/15 | 3/3 | 7/10 | 4/5 | 11/20 | 17/22 | 12/16 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Setmelanotide 0.5 mg (Double-blind Randomized Treatment) (N=4) | Setmelanotide 1.5 mg (Double-blind Randomized Treatment) (N=13) | Setmelanotide 2.5 mg (Double-blind Randomized Treatment) (N=8) | Placebo (Double-blind Randomized Treatment) (N=15) | Setmelanotide 0.5 mg (Randomized Withdrawal Period) (N=3) | Setmelanotide 1.5 mg (Randomized Withdrawal Period) (N=10) | Setmelanotide 2.5 mg (Randomized Withdrawal Period) (N=5) | Placebo (Randomized Withdrawal Period) (N=20) | Setmelanotide 1.5 mg (Open-Label Extension) (N=22) | Setmelanotide 2.5 mg (Open-Label Extension) (N=16) | Placebo (Open-Label Extension) (N=1)
Injection site erythema (General disorders) | 3 | 5 | 4 | 6 | 2 | 4 | 4 | 4 | 8 | 6 | 0
Injection site induration (General disorders) | 2 | 4 | 2 | 3 | 2 | 2 | 0 | 4 | 6 | 6 | 0
Injection site oedema (General disorders) | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 6 | 2 | 0
Injection site bruising (General disorders) | 3 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 5 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Injection site pruritus (General disorders) | 1 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discolouration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site nodule (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site erosion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erection increased (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spontaneous penile erection (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital disorder female (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tearfulness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Libido increased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pigmentation lip (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2016-01-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT02311673/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT02311673/SAP_001.pdf